CLINICAL TRIAL: NCT04201899
Title: Hypophosphatemia in the ICU - A One-day Point Prevalence Survey
Brief Title: HYPOPhosphatemia in the Intensive Care: A One-day Point Prevalence Survey
Acronym: HYPO-P-ICU
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Principal Investigator, Mette M Berger, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Other Study IDs: CER2019-02343; 2019-021-406 (Other: Erasme University, Brussels, Belgium)
Record Dates: First submitted 2019-12-14; First posted 2019-12-17 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Critically Ill
Keywords: Phosphate
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: No intervention - pure observation — Phosphate administration (yes or no)

SUMMARY:
The point prevalence survey aims at defining the until now unknown real prevalence of hypophosphatemia (defined as blood phosphate value < 0.8 mmol/l) in international critical care settings

DETAILED DESCRIPTION:
The survey will be conducted on one single day in each centre (D-day), within a week defined by the project coordinator (International PI). On D-Day, the local investigators will be asked

1. to complete questions aiming at describing their ICU (number of beds, number of patients present on D-Day, type medical/surgical/other, local phosphate reference value, presence of an hypophosphatemia treatment protocol in the ICU and route of phosphate delivery in case of hypophosphatemia)
2. to indicate how many patients had a blood phosphate <0.08 mmol/l, for each patient with hypophosphatemia, to record the exact lowest value on D-Day, and to record age, number of days in ICU on D-Day, presence (or not) of artificial nutrition and continuous renal replacement therapy, if any phosphate administration is ongoing Data will be recorded in and electronic Case Report Form (e-CRF) in REDCap, and analysed with descriptive statistics No outcome data will be recorded (pure point-prevalence) There is no intervention

ELIGIBILITY:
Inclusion Criteria: blood phosphate value < 0.8 mmol -

Exclusion Criteria: Blood phosphate value >0.8 mmol/l

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients: adults and children
Sampling Method: Non-Probability Sample
Enrollment: 890 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of hypophosphatemia | 1 day
  Blood value < 0.8 mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Mette M BERGER, MD PhD, Principal Investigator — Lausanne University Hospital, Lausanne, Switzerland
Locations (4):
- Tartu University Hospital, Tartu, Estonia
- Hôpital Pasteur 2, Nice, France
- Switzerland (2):
  - Lausanne University Hospital, Lausanne, Canton of Vaud
  - Hôpital de Nyon, Nyon

IPD SHARING:
Plan to Share IPD: No
Data will be collected in central REDCap database. No individual patient data will be made available

REFERENCES:
- [Derived] Berger MM, Appelberg O, Reintam-Blaser A, Ichai C, Joannes-Boyau O, Casaer M, Schaller SJ, Gunst J, Starkopf J; ESICM-MEN section. Prevalence of hypophosphatemia in the ICU - Results of an international one-day point prevalence survey. Clin Nutr. 2021 May;40(5):3615-3621. doi: 10.1016/j.clnu.2020.12.017. Epub 2020 Dec 29. PMID 33454128